CLINICAL TRIAL: NCT02704650
Title: Identification and Characterization of Ovarian Cancer and Endometrial Cancer Specific Biomarkers in Vaginal Fluids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Gina-Life Diagnostics ltd. (Industry)
Responsible Party: Principal Investigator, Shachar Finci, Principal Investigator, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Shachar-1
Record Dates: First submitted 2016-02-11; First posted 2016-03-10 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Cancer of Ovary
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal fluid of healthy patient (Experimental): vaginal fluid sample from healthy patients
  Interventions: Procedure: fluid sample
- Vaginal fluid of ovary cancer patients (Experimental): vaginal fluid sample from patients with ovary cancer
  Interventions: Procedure: fluid sample

INTERVENTIONS:
Procedure: fluid sample — taking a vaginal fluid sample

SUMMARY:
The purpose of this study is to:

1. Identification and characterization of ovarian carcinoma well-known biomarkers, carcinoma antigen 125 (CA125) and Human epididymis protein 4 (HE4) and other potential biomarkers in vaginal fluids obtained from ovarian cancer patients.
2. Quantification and calibration of identified biomarkers in vaginal discharge collected from ovarian cancer patients in comparisons to samples collected from healthy volunteers.
3. Comparison analysis of biomarkers levels in vaginal fluids vs. serum.
4. Quantification and calibration of identified biomarkers in vaginal discharge collected from ovarian cancer patients diagnosed in various stages.

DETAILED DESCRIPTION:
Initially, twenty vaginal fluid samples will be collected from ovarian cancer patients diagnosed with epithelial ovarian carcinoma at advanced diagnosis stage.

The samples will be used to identify specific biomarkers as describe above. Biomarkers levels will be calibrated compared to their vaginal fluids obtained from healthy volunteers. In addition, five milliliters of venous blood will be collected from same patients in order to compare biomarkers vaginal fluids levels vs serum levels. All patients will sign a consent form which approve that their vaginal fluid samples will be utilized for research according to Helsinki approval.

At the second phase of the research, additional twenty vaginal fluids samples will be collected from patients diagnosed at different stages (five samples from each of main stages 1-4). Sample will be used to calibrate biomarkers levels in various diagnosis stages and will be compare to serum levels from venous blood samples which will be also collected from the same patients.

All patients will sign a consent form following explanation on research goals. Patient will be notified that participation in this research will have no implication on medical treatment plan.

Note that in all research phases there will be no returning of samples to the patients, all identification and characterization procedures will be performed in vitro for research properties only.

Methodology

* Collecting vaginal fluids samples from ovarian cancer patients. Vaginal fluids (at least 400µl, the investigators wish to have 1000 µl) will be collected during surgery or during routine physical examination using specific applicator/cotton swab/syringe. Samples will be shipped to GinaLife Diagnostics laboratory for analysis. In addition, on the day of vaginal fluids collection 5 ml of peripheral blood samples will be drawn from each volunteer.
* Analyzing specific biomarkers in samples. Vaginal fluids will be analyzed using commercial enzyme-linked immunosorbent assay (ELISA) kits to determine the presence and the concentrations of various proteins. In addition, western blot analysis will be used in order to confirm ELISA assay results. Specific nucleic acid will be determine using common molecular methods such as Reverse transcription polymerase chain reaction (RT-PCR) etc.
* Data analysis

ELIGIBILITY:
Inclusion Criteria:

* Ovarian carcinoma (in the "disease" arm)

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The difference in the levels of the Human Epididymis Protein 4 (HE4) measured between healthy patients and ovary cancer patients. Measuring units will be pmol/L. | 1 year
The difference in the levels of the glycoprotein CA-125 between healthy patients and ovary cancer patients. The measuring units will be U/mL. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shachar Finci, MD, Principal Investigator — Shaare Zedek Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orfanelli T, Jayaram A, Doulaveris G, Forney LJ, Ledger WJ, Witkin SS. Human epididymis protein 4 and secretory leukocyte protease inhibitor in vaginal fluid: relation to vaginal components and bacterial composition. Reprod Sci. 2014 Apr;21(4):538-42. doi: 10.1177/1933719113503416. Epub 2013 Sep 10. PMID 24023032
- [Result] Montagnana M, Lippi G, Ruzzenente O, Bresciani V, Danese E, Scevarolli S, Salvagno GL, Giudici S, Franchi M, Guidi GC. The utility of serum human epididymis protein 4 (HE4) in patients with a pelvic mass. J Clin Lab Anal. 2009;23(5):331-5. doi: 10.1002/jcla.20340. PMID 19774626
- [Result] Drapkin R, von Horsten HH, Lin Y, Mok SC, Crum CP, Welch WR, Hecht JL. Human epididymis protein 4 (HE4) is a secreted glycoprotein that is overexpressed by serous and endometrioid ovarian carcinomas. Cancer Res. 2005 Mar 15;65(6):2162-9. doi: 10.1158/0008-5472.CAN-04-3924. PMID 15781627
- [Result] Kim A, Ueda Y, Naka T, Enomoto T. Therapeutic strategies in epithelial ovarian cancer. J Exp Clin Cancer Res. 2012 Feb 13;31(1):14. doi: 10.1186/1756-9966-31-14. PMID 22330607